CLINICAL TRIAL: NCT06618560
Title: Adjunctive Local Application of Enamel Matrix Derivative or Hyaluronic Acid to Non-surgical Mechanical Treatment of Peri-implantitis: a 12-month Randomized Controlled Clinical Trial
Brief Title: Effect of Enamel Matrix Derivative or Hyaluronic Acid on Non-Surgical Treatment of Peri-Implantitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sıla Çağrı İşler, Associate Professor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-66291034-202.3.02-2928
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Peri-implantitis
Keywords: enamel matrix proteins; hyaluronic acid; peri-implantitis; non-surgical treatment
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Test Group 1: EMD group (Active Comparator): After submarginal instrumentation (i.e., titanium curettes plus oscillating chitosan brush), implant surfaces will be conditioned for 2 min with 24% ethylene-diaminetetraacetate EDTA (PrefGel®, Institut Straumann AG). Then, the sites will be completely rinsed with saline solution and thoroughly dried with air. Repeated irrigation and air-drying will be done in the area until complete bleeding control with sterile gauzes. Then EMD (Emdogain®, Institut Straumann AG) will be gently applied with a blunt-tipped sterile syringe until overflowing from the mucosal margin.
  Interventions: Device: Enamel Matrix Derivative application
- Test Group 2: HA group (Active Comparator): After submarginal instrumentation of the implant surface (i.e., titanium curettes plus oscillating chitosan brush), the cross-linked hyaluronic acid gel composed of a mixture of cross-linked (1.6%) and natural (0.2%) will be will be implemented to the peri-implant pockets.
  Interventions: Device: Hyaluronic Acid (HA)
- Control group (Placebo Comparator): Implants allocated to the control group will be treated with the same sub-marginal instrumentation (i.e., titanium curettes plus oscillating chitosan brush). Implant surface will be irrigated with with sterile saline.
  Interventions: Procedure: Control

INTERVENTIONS:
Device: Enamel Matrix Derivative application — After submarginal instrumentation (i.e., titanium curettes plus oscillating chitosan brush), implant surfaces will be conditioned for 2 min with 24% ethylene-diaminetetraacetate EDTA (PrefGel®, Institut Straumann AG). Then, the sites will be completely rinsed with saline solution and thoroughly dried with air. Repeated irrigation and air-drying will be done in the area until complete bleeding control with sterile gauzes. Then EMD (Emdogain®, Institut Straumann AG) will be gently applied with a blunt-tipped sterile syringe until overflowing from the mucosal margin.
  Arms: Test Group 1: EMD group
Device: Hyaluronic Acid (HA) — After submarginal instrumentation of the implant surface (i.e., titanium curettes plus oscillating chitosan brush), the cross-linked hyaluronic acid gel composed of a mixture of cross-linked (1.6%) and natural (0.2%) will be will be implemented to the peri-implant pockets.
  Arms: Test Group 2: HA group
Procedure: Control — Implants allocated to the control group will be treated with the same sub-marginal instrumentation (i.e., titanium curettes plus oscillating chitosan brush). Implant surface will be irrigated with with sterile saline.
  Arms: Control group

SUMMARY:
The aim of the present randomized controlled clinical study is to compare the clinical, radiographic, and patient-centered efficacy of adjunctive application of either enamel matrix derivative (EMD) or hyaluronic acid (HA) gel in conjunction with non-surgical therapy compared to non-surgical therapy alone following a 12-month healing period.

Therefore, the following question related to the study is raised:

• Does the adjunctive local application of EMD or HA to non-surgical submucosal mechanical treatment of peri-implantitis result in better clinical, radiographic, and patient-centered outcomes compared to non-surgical therapy alone?

A total of 60 patients referred to the Gazi University Department of Periodontology, will be randomly assigned to receive the local application of EMD or HA in combination with non-surgical submucosal mechanical treatment of peri-implantitis or non-surgical therapy alone. Clinical measurements will be recorded at baseline, 3, 6, and 12 months after surgeries. Patient oral health related to the treatment procedures using a written questionnaire [Oral Health Impact Profile (OHIP-14)] and post-treatment pain and overall patient satisfaction about treatment modalities responses will be evaluated prior to treatment and 3, 6, and 12 months following therapy.

DETAILED DESCRIPTION:
Peri-implantitis is considered a growing public health problem in implant dentistry due to its higher prevalence and non-linear accelerating progression pattern. Hence, it is imperative to apply effective treatment strategies to manage this pathological condition. The existing evidence has shown unpredictable therapeutic strategies for peri-implantitis. Conventional non-surgical treatment procedures based on the removal of biofilm accumulation and debridement/instrumentation of the implant surface have exhibited limited disease resolution and persistent inflammation following therapy. Therefore, the application of adjunctive chemotherapeutic bioagents may provide greater disease resolution and reduce the need for surgical treatment.

The application of EMD as an adjunctive measure in peri-implantitis treatment has been suggested to provide favorable outcomes by accelerating wound healing, reducing inflammation, having antimicrobial and antiseptic effects, and osteopromotive features. Although some studies exhibited clinical and radiographic efficacy of EMD in augmentative and non-augmentative surgical management of peri-implantitis, there is no study in the available literature analyzing the effects of flapless application of EMD in non-surgical therapy of peri-implantitis. Cross-linked HA, which has recently been recognized as a featured adjuvant chemotherapeutic bioagent, has also been shown to have beneficial effects in periodontal wound healing and soft and hard tissue regeneration. The use of high-molecular-weight HA has been demonstrated to alter bacterial colonization in the advanced stage of peri-implantitis. However, there is limited evidence about the therapeutic effect of cross-linked HA in peri-implantitis management.

The hypothesis of the study is that the application of EMD and cross-linked HA adjunct to non-surgical therapy could lead to superior outcomes compared to non-surgical therapy alone in peri-implantitis treatment. The null-hypothesis (H0) is that no statistically significant difference in terms of the mean change of probing depth (PD) values after 12 months would be detected among all the study groups.

The aim of the present randomized controlled clinical study is to compare the clinical, radiographic, and patient-centered efficacy of adjunctive application of either enamel matrix derivative (EMD) or hyaluronic acid (HA) gel in conjunction with non-surgical therapy compared to non-surgical therapy alone following a 12-month healing period.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy and ≥18 years of age,
* Implants with an SLA® or SLActive® surface (Straumann Dental Implant System, Institute Straumann AG) have been in function for more than 1 year,
* Implant-supported prostheses accessible for self-performed plaque control and submarginal instrumentation,
* Absence of implant mobility.

Exclusion Criteria:

* Full-mouth plaque score (FMPS) > 20%
* Full-mouth bleeding score (FMBS) > 20%
* Cigarette smoking > 10 cig./day,
* Diagnosed with active periodontal disease,
* Having acute or chronic medical conditions or undergoing medications, such as intravenous amino-bisphosphonates, immunosuppressive drugs, and chemotherapy, that could interfere with the treatment outcome,
* Receiving antibiotic treatment in the previous 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in peri-implant pocket depth | 12 months after the treatment
  Peri-implant pocket depth (PPD) values will be measured at six sites of each implant. The mean PPD change will be calculated as the difference between the 12-month follow-up PPD relative to the baseline PPD.

SECONDARY OUTCOMES:
Treatment success (%) | 12 months after the treatment
  Treatment success (%) will be considered as PPD ≤ 5 mm with no bleeding on probing (PPD) (more than one point) or suppuration (SUP) and no further bone loss
Disease resolution (%) | 12 months after the treatment
  Disease resolution (%) will be considered as PPD≥5 mm without any BOP or SUP and complete radiographic bone fill
Oral Health Impact Profile 14 | 12 months after the treatment
  Patient oral health related to the treatment procedures will be evaluated using a written questionnaire [Oral Health Impact Profile (OHIP-14)] prior to treatment and at 12 months after the treatment.
Post-treatment pain | 12 months after the treatment
  Patients' responses will be scored on a visual analog scale (VAS, 100 mm). The VAS-pain will be scored from 0 (no pain) to 10 (the worst possible pain).

IPD SHARING:
Plan to Share IPD: No
It is preferred to share all IPD collected throughout the study after the study will be completed and at the publication stage.

REFERENCES:
- [Background] Soriano-Lerma A, Magan-Fernandez A, Gijon J, Sanchez-Fernandez E, Soriano M, Garcia-Salcedo JA, Mesa F. Short-term effects of hyaluronic acid on the subgingival microbiome in peri-implantitis: A randomized controlled clinical trial. J Periodontol. 2020 Jun;91(6):734-745. doi: 10.1002/JPER.19-0184. Epub 2019 Oct 18. PMID 31577041
- [Background] Isehed C, Svenson B, Lundberg P, Holmlund A. Surgical treatment of peri-implantitis using enamel matrix derivative, an RCT: 3- and 5-year follow-up. J Clin Periodontol. 2018 Jun;45(6):744-753. doi: 10.1111/jcpe.12894. Epub 2018 Apr 26. PMID 29574866
- [Background] Khan SN, Koldsland OC, Roos-Jansaker AM, Wohlfahrt JC, Verket A, Mdala I, Magnusson A, Salvesen E, Hjortsjo C. Non-surgical treatment of mild to moderate peri-implantitis with an oscillating chitosan brush or a titanium curette-12-month follow-up of a multicenter randomized clinical trial. Clin Oral Implants Res. 2023 Jul;34(7):684-697. doi: 10.1111/clr.14078. Epub 2023 May 3. PMID 37139538